CLINICAL TRIAL: NCT00467207
Title: Intensive Strength Training in Children With Cerebral Palsy - Effect on Hand Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/1553
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BoNT A (Active Comparator): Botulinum toxin A injections in muscles of the arm (biceps brachii and brachialis)
  Interventions: Drug: Botulinum Toxin A
- Resistance training (Experimental): 8 weeks resistance training
  Interventions: Drug: Botulinum Toxin A; Behavioral: Resistance training

INTERVENTIONS:
Drug: Botulinum Toxin A
  Other Names: Botox; BoNT A
Behavioral: Resistance training
  Other Names: Strength training
  Arms: Resistance training

SUMMARY:
The objective of this study is to gain more knowledge about the association between muscle weakness, spasticity and motor control in children with cerebral palsy, and its relationship to hand function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed spastic hemiplegic or diplegic cerebral palsy, reduced handfunction.
* Indication for treatment with Botulinum Toxin A
* Score 3 on House Classification of Upper-Extremity Functional Use
* Score 3 or better on Manual Ability Classification System

Exclusion Criteria:

* surgery within the last two years
* Treatment with Botulinum Toxin within the last six months

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torarin I Lamvik, md, Study Chair — St. Olavs Hospital; Karin Roeleveld, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Elvrum AK, Braendvik SM, Saether R, Lamvik T, Vereijken B, Roeleveld K. Effectiveness of resistance training in combination with botulinum toxin-A on hand and arm use in children with cerebral palsy: a pre-post intervention study. BMC Pediatr. 2012 Jul 2;12:91. doi: 10.1186/1471-2431-12-91. PMID 22747635
- [Result] Braendvik SM, Elvrum AK, Vereijken B, Roeleveld K. Relationship between neuromuscular body functions and upper extremity activity in children with cerebral palsy. Dev Med Child Neurol. 2010 Feb;52(2):e29-34. doi: 10.1111/j.1469-8749.2009.03490.x. Epub 2009 Oct 7. PMID 19811515
- [Result] Braendvik SM, Roeleveld K. The role of co-activation in strength and force modulation in the elbow of children with unilateral cerebral palsy. J Electromyogr Kinesiol. 2012 Feb;22(1):137-44. doi: 10.1016/j.jelekin.2011.10.002. Epub 2011 Nov 8. PMID 22071153